CLINICAL TRIAL: NCT05348785
Title: A Phase 2b, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Determine the Efficacy and Safety of BIIB122 in Participants With Parkinson's Disease
Brief Title: A Study to Learn About the Safety of BIIB122 Tablets and Whether They Can Slow the Worsening of Early-Stage Parkinson's Disease in Adults Between the Ages of 30 and 80
Acronym: LUMA
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Collaborators: Denali Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 283PD201; 2023-505645-12 (Other: EU CT Number)
Record Dates: First submitted 2022-04-04; First posted 2022-04-27 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Parkinson Disease
Keywords: Early-stage Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — DNL151

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BIIB122 225 mg (Experimental): Participants will receive BIIB122, 225 mg tablets, by mouth, once daily (QD) for up to a minimum of 48 weeks and a maximum of 144 weeks.
  Participants who received BIIB122 and completed the ET visit of study 283PD302 (NCT05418673) will continue to receive BIIB122, 225 mg tablets, by mouth, QD for up to a minimum of 48 weeks and a maximum of 144 weeks.
  Interventions: Drug: BIIB122
- BIIB122 Matching Placebo (Placebo Comparator): Participants will receive BIIB122 matching placebo tablets, by mouth, QD for up to a minimum of 48 weeks and a maximum of 144 weeks.
  Participants who received placebo and completed the ET visit of study 283PD302 (NCT05418673) will continue to receive BIIB122 matching placebo tablets, by mouth, QD for up to a minimum of 48 weeks and a maximum of 144 weeks.
  Interventions: Drug: BIIB122-Matching Placebo

INTERVENTIONS:
Drug: BIIB122 — Administered as specified in the treatment arm
  Other Names: DNL151
  Arms: BIIB122 225 mg
Drug: BIIB122-Matching Placebo — Administered as specified in the treatment arm
  Arms: BIIB122 Matching Placebo

SUMMARY:
In this study, researchers will learn more about BIIB122 in participants with early-stage Parkinson's disease (PD). The study will include adults aged 30 to 80 who were diagnosed with PD within 2 years of starting the study.

The main objective of the study is to learn about the effect BIIB122 has on slowing down the worsening of PD symptoms. The main question researchers want to answer is:

- How long does it take for PD symptoms to worsen during BIIB122 treatment?

Researchers will answer this and other questions by measuring the symptoms of PD over time using a variety of scoring tools. These include the Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) and the modified Schwab and England Activities of Daily Living Scale (mSE-ADL).

The MDS-UPDRS is used to measure symptoms of PD. It has 4 parts: Part I, II, III, and IV. Each part measures different aspects of motor and non-motor symptoms. The mSE-ADL measures a participant's ability to perform daily activities or personal chores.

Researchers will also learn more about the safety of BIIB122. They will check participants for adverse events. Adverse events are unwanted health problems that may or may not be caused by the study drug.

The study will be done as follows:

* Participants will be randomly assigned to take either BIIBB122 or placebo. A placebo looks like the study drug but contains no real medicine.
* Neither the researchers nor the participants will know if the participants are receiving BIIB122 or placebo.
* Participants will take BIIB122 or placebo tablets by mouth once a day.
* The treatment period for each participant will last between 48 and 144 weeks.
* There will be a safety follow-up period for 2 weeks after the last dose of BIIB122.
* In total, participants will have up to 29 study visits.
* Participants will stay in the study for at least 1 year, up to about 3 years.

DETAILED DESCRIPTION:
BIIB122 is an investigational central nervous system-penetrant small molecule inhibitor of leucine-rich repeat kinase 2 (LRRK2). Participants who completed the early termination (ET) visit of the study 283PD302 (NCT05418673) would be eligible for screening of this study and if enrolled, these participants are not eligible for the sub studies of 283PD201.

ELIGIBILITY:
Key Inclusion Criteria:

* Clinical diagnosis of PD meeting the Movement Disorder Society Clinical Diagnostic Criteria within 2 years of the Screening Visit, inclusive, and at least 30 years of age at the time of diagnosis
* Modified Hoehn and Yahr scale stages 1 to 2 (in OFF state), inclusive, at screening
* MDS-UPDRS Parts II and III (in OFF state) combined score less than or equal to (≤)50 at screening

Key Exclusion Criteria:

* Clinically significant neurological disorder other than PD, including but not limited to stroke, dementia, or seizure, within 5 years of screening visit, in the opinion of the Investigator
* Clinical evidence of atypical parkinsonism (e.g., multiple-system atrophy or progressive supranuclear palsy) or evidence of drug-induced parkinsonism.
* Montreal Cognitive Assessment (MoCA) score <24 at the screening visit.

NOTE: Other protocol-defined Inclusion/Exclusion criteria may apply.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Actual)
Dates: Start 2022-04-19 (Actual); Primary Completion 2026-02-25 (Estimated); Study Completion 2026-03-09 (Estimated)

PRIMARY OUTCOMES:
Time to Confirmed Worsening in Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Parts II and III Combined Score Over the Treatment Period | Up to Week 144
  Time to confirmed worsening is defined as a worsening event sustained over 2 consecutive assessments. MDS-UPDRS is a multimodal scale assessing impairment and disability consisting of 4 parts. Part II assesses motor experiences of daily living (Range 0-52). It contains 13 questions which are to be completed by the participant. Part III assesses the motor signs of PD and is administered by the rater (Range 0-132). Part III contains 33 scores based on 18 items. For each question a numeric score is assigned between 0-4, where 0 = Normal, 1 = Slight, 2 = Mild, 3 = Moderate, 4 = Severe. MDS-UPDRS Part II and III combined score equals the sum of Parts II and III (Range 0-184). A higher score indicates more severe symptoms of PD.

SECONDARY OUTCOMES:
Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Up to Week 144
  An AE is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. An SAE is any untoward medical occurrence that at any dose results in death; in the view of the investigator, places the participant at immediate risk of death (a life-threatening event); requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; results in a congenital anomaly/birth defect or is a medically important event.
Time to Confirmed Worsening in MDS-UPDRS Part II Score Over the Treatment Period | Up to a minimum of 48 weeks and a maximum of 144 weeks
  Time to confirmed worsening is defined as a worsening event sustained over 2 consecutive assessments. MDS-UPDRS is a multimodal scale assessing impairment and disability consisting of 4 parts. Part II assesses motor experiences of daily living (Range 0-52). It contains 13 questions which are to be completed by the participant. For each question a numeric score is assigned between 0-4, where 0 = Normal, 1 = Slight, 2 = Mild, 3 = Moderate, 4 = Severe. A higher score indicates more severe symptoms of PD.
Change From Baseline in MDS-UPDRS Parts II and III Combined Score | From Baseline up to Week 48
  MDS-UPDRS is a multimodal scale assessing impairment and disability consisting of 4 parts. Part II assesses motor experiences of daily living (Range 0-52). It contains 13 questions which are to be completed by the participant. For each question a numeric score is assigned between 0-4, where 0 = Normal, 1 = Slight, 2 = Mild, 3 = Moderate, 4 = Severe. A higher score indicates more severe symptoms of PD. Part III assesses the motor signs of PD and is administered by the rater (Range 0-132). Part III contains 33 scores based on 18 items. For each question a numeric score is assigned between 0-4, where 0 = Normal, 1 = Slight, 2 = Mild, 3 = Moderate, 4 = Severe. MDS-UPDRS Parts II and III combined score equals the sum of Part II and III (Range 0-184). A higher score indicates more severe symptoms of PD.
Time to Confirmed Worsening in Modified Schwab and England Activities of Daily Living Scale (mSE-ADL) Over the Treatment Period | Up to a minimum of 48 weeks and a maximum of 144 weeks
  Time to confirmed worsening is defined as a worsening event sustained over 2 consecutive assessments. The mSE-ADL scale reflects the speed, ease, and independence with which an individual performs daily activities or personal chores with 100% indicating total independence, falling to 0%, which indicates a state of complete dependence. The individual is asked to rate his or her function using an 11-point scale (10% increments), from 100% (completely independent; able to do all chores without slowness, difficulty, or impairment; essentially normal; unaware of any difficulty) to 0% (vegetative functions such as swallowing, bladder and bowels are not functioning; bedridden). The lower the score, the worse the functional status.
Change From Baseline in MDS-UPDRS Parts I, II, and III Combined Score | From Baseline up to Week 48
  MDS-UPDRS is a multimodal scale assessing impairment and disability consisting of 4 parts. Part I assesses non-motor experiences of daily living and has 2 components (Range 0-52). Part IA contains 6 questions and is assessed by the examiner (Range 0-24). Part IB contains 7 questions on non-motor experiences of daily living which are to be completed by the participant (Range 0-28). Part II assesses motor experiences of daily living (Range 0-52). It contains 13 questions which are to be completed by the participant. Part III assesses the motor signs of PD and is administered by the rater (Range 0-132). Part III contains 33 scores based on 18 items. For each question a numeric score is assigned between 0-4, where 0 = Normal, 1 = Slight, 2 = Mild, 3 = Moderate, 4 = Severe. MDS-UPDRS total score equals the sum of Parts I, II, and III (Range 0-236). A higher score indicates more severe symptoms of PD.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (113):
- United States (33):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Banner Sun Health Research Institute, Sun City, Arizona
  - University of Southern California, Los Angeles, California
  - Cedars Sinai, Los Angeles, California
  - SC3 Research Group Inc., Pasadena, California
  - University of California San Francisco (UCSF), San Francisco, California
  - University of Colorado, Aurora, Colorado
  - CenExel Rocky Mountain Clinical Research, Englewood, Colorado
  - Invicro, New Haven, Connecticut
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - University of Miami, Miami, Florida
  - Adventist Health System/Sunbelt, Inc., Orlando, Florida
  - USF Health Byrd Institute, Tampa, Florida
  - Hawaii Pacific Neuroscience, LLC, Honolulu, Hawaii
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Kansas Medical Center Research Institute, Inc., Kansas City, Kansas
  - Boston University Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Quest Research Institute, Farmington Hills, Michigan
  - Mount Sinai Beth Israel, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - Duke Movement Disorders Clinic, Durham, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - UPHS, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Neurology Clinic, PC, Cordova, Tennessee
  - The Methodist Hospital Research Institute, Houston, Texas
  - Central Texas Neurology Consultants, Round Rock, Texas
  - Virginia Commonwealth University Department of Neurology, Richmond, Virginia
  - Evergreen Hospital Medical Center, Kirkland, Washington
  - Inland Northwest Research, Spokane, Washington
- Austria (2):
  - Medizinische Universität, Innsbruck, Tyrol
  - Klinik Ottakring, Vienna
- Canada (5):
  - University of Calgary, Calgary, Alberta
  - True North Clinical Research, Halifax, Nova Scotia
  - Toronto Western Hospital, Toronto, Ontario
  - CHUM Centre de Recherche, Montreal, Quebec
  - Montreal Neurological Institute, Montreal, Quebec
- China (4):
  - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Second Affiliated Hospital of Soochow University, Jiangsu, Jiangsu
  - West China Hospital, Sichuan University, Chengdu, Sichuan
- France (9):
  - Hôpital de la Timone, Marseille, Bouches-du-Rhône
  - Hopital Purpan, Toulouse, Haute Garonne
  - Hopital Gui de Chauliac, Montpellier, Herault
  - CHU Rennes - Hopital Pontchaillou, Rennes, Ille Et Vilaine
  - CHU Nantes - Hopital Nord Laën, Loire-Atlantique, Loire-Atlantique
  - CHU Clermont Ferrand - Hopital Gabriel Montpied, Clermont-Ferrand, Puy De Dome
  - Centre Hospitalier Universitaire de Lyon-Hospices Civils de Lyon-Hopital Pierre Wertheimer, Bron, Rhone
  - Groupe Hospitalier Pitie-Salpetriere, Paris
  - Hopital Henri Mondor, Paris
- Germany (12):
  - Universitaetsklinikum Tuebingen, Tübingen, Baden-Wurttemberg
  - Universitaetsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Klinikum der Universität München, Munich, Bavaria
  - Klinikum rechts der Isar der TU Muenchen, Munich, Bavaria
  - Universitaetsklinikum Wuerzburg, Würzburg, Bavaria
  - Paracelsus-Elena-Klinik Kassel, Kassel, Hesse
  - Philipps University of Marburg, Marburg, Hesse
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Katholisches Klinikum Bochum gGmbH, Bochum, North Rhine-Westphalia
  - Universitaetsklinikum Duesseldorf AoeR, Düsseldorf, North Rhine-Westphalia
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Dresden, Saxony
  - Universitaetsklinikum Schleswig-Holstein - Campus Luebeck, Lübeck, Schleswig-Holstein
- Israel (3):
  - Rabin Medical Center, Petah Tikva
  - Center Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (10):
  - I.R.C.C.S. Neuromed, Diego, Centonze
  - IRCCS-Institute of Neurological Sciences of Bologna, Bologna
  - Azienda Ospedaliera Spedali, Brescia
  - Azienda Ospedaliero Universitaria Policlinico 'Gaspare Rodolico - San Marco' (Presidio G. Rodolico), Catania
  - Ospedale Clinicizzato SS. Annu, Chieti
  - Fondazione, Milan
  - Ospedale San Raffaele, Milan
  - AOU Luigi Vanvitelli, Napoli
  - AO Universitaria Pisana, Pisa
  - IRCCS San Raffaele Pisana, Roma
- Japan (6):
  - Okinawa Prefectural Nanbu, Haeburu, Okinawa
  - Tazuke-kofukai Medical Research Institute Kitano Hospital, Osaka, Osaka
  - NHO Asahikawa Medical Center, Asahikawa-shi
  - Himeji Central, Himeji-shi
  - Sendai Nishitaga National Hospital, Sendai
  - Juntendo University, Tokyo
- Netherlands (3):
  - Brain Research Center Amsterdam, Amsterdam
  - Radboudumc, Nijmegen
  - Brain Research Center Zwolle B.V., Zwolle
- Poland (6):
  - Instytut Zdrowia dr Boczarska-Jedynak sp.z.o.o, Sp.K, Oświęcim, Katowice
  - NeuroProtect Sp. z o.o., Warsaw, Masovian Voivodeship
  - Centrum Medyczne Neuromed, Bydgoszcz
  - Nzoz Novo-Med, Katowice
  - INSULA Centrum Badan Klinicznych, Warsaw
  - MD Clinic Praga, Warsaw
- Spain (11):
  - Hospital General de Catalunya, Sant Cugat del Vallès, Barcelona
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitario Marques, Santanda, Santanda
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital de Cruces, Barakaldo
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Policlinica Gipuzkoa, Donostia / San Sebastian
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
- United Kingdom (9):
  - University Hospitals Plymouth, Plymouth, Devon
  - Re:Cognition Health Ltd (London), London, Greater London
  - Charing Cross Hospital, London, Greater London
  - The National Hospital for Neurology & Neurosurgery, London, Greater London
  - Salford Royal NHS Foundation Trust, Salford, Greater Manchester
  - NeuroClin Limited, Motherwell, Strathclyde
  - Newcastle University, Newcastle upon Tyne, Tyne and Wear
  - Re:Cognition Health - Birmingham, Birmingham, West Midlands
  - Ninewells Hospital, Dundee

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

REFERENCES:
- [Derived] Joshi D, Kulkarni M, Parekh P, Shah S, Greig NH, Acharya S. Targeting protein kinases in Parkinson's disease: the emerging role of phytoconstituents. Nutr Neurosci. 2025 Dec;28(12):1532-1563. doi: 10.1080/1028415X.2025.2531356. Epub 2025 Jul 18. PMID 40680102